CLINICAL TRIAL: NCT05801263
Title: ctDNA Methylation Testing for Detecting Epithelial Ovarian Cancer: A Prospective Multicenter Cohort Study (OVAMethy Study)
Brief Title: ctDNA Methylation for Epithelial Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: OVAMethy
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Epithelial Ovarian Cancer; Circulating Tumor DNA; DNA Methylation; Non-invasive Diagnosis; CA125; Human Epididymis Protein 4; Imaging Evaluation; Survival Prognosis
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma circulating tumor DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CDO1 and HOXA9 methylation assay — CDO1 and HOXA9 methylation assay in plasma circulating tumor cells

SUMMARY:
Ovarian cancer is one of the most dangerous and predominant gynecological cancers, with a high cancer-related mortality rate in women. However, current testing methods are still limited, and if detected early, patients have a five-year survival rate of 92%. Therefore, early diagnosis and detection are crucial for diagnosing and treating ovarian cancer. According to the results of the researchers' previous research, it has been found that CDO1 and HOXA9 genes are hypermethylated in ovarian cancer, and the expression of free DNA methylation in plasma can be used as one of the biomarkers for detection. In a single-center retrospective/prospective study, it has been demonstrated that the detection of CDO1 and HOXA9 methylation levels based on cell-free DNA in blood and comparison with ovarian pathology results can achieve >80% sensitivity and specificity. To further explore the application of methylation detection technology in ovarian cancer, the application value of non-invasive diagnosis and prognosis follow-up will be explored to clarify the clinical application value of DNA methylation for early detection of ovarian cancer in the real world. The investigators will conduct a prospective multi-center cohort study, referred to as the OVAMethy study, which will involve more than ten research centers and is expected to recruit more than 5,000 clinical subjects to test the methylation detection kit and histopathology further, ROMA index and imaging results, and sensitivity and specificity technical performance parameters.

DETAILED DESCRIPTION:
In this study, cell-free DNA will be extracted from the blood of outpatient opportunistic screening subjects, the methylation status of genes will be measured, and the test results will be obtained. Histological sampling was performed by current clinical practice in patients with clinical manifestations and corresponding examinations (e.g., abnormal uterine bleeding, ovarian mass/cyst on ultrasound, elevated tumor markers) suggesting ovarian lesions. Accuracy of screening for ovarian cancer based on histopathological analysis of blood ctDNA methylation. A 12-month clinical follow-up of women with DNA methylation at risk for ovarian cancer, including symptom analysis, physical examination, imaging studies (ultrasound, CT, or MRI), surgery or (biopsy) pathology, and tumors such as ROMA Marker determination. Collect 5ml of blood for methylation testing before treatment. For the hospital for treatment follow-up, the scheme for collecting patient information includes basic data (birthday, medical record number, height, weight, etc.), symptom analysis, physical examination, imaging examination (ultrasound, CT or MRI), surgery or (biopsy) pathology, Determination of tumor markers such as ROMA, as well as the use of main therapeutic drugs and courses of treatment, time to recurrence, re-treatment plan and course of treatment, time of death (such as those who died during the study), etc. Blood was collected for methylation detection. The 5ml blood collection points were (1). Before treatment (surgery/chemoradiotherapy/immunotherapy); (2). Follow-up visit one month after treatment; (3). Follow-up 3rd and 6th after treatment, 9, and 12 months, and complete follow-up cases and specimen collection before March 24, 2024.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient routine follow-up population
* Age is greater than or equal to 18 years
* Not receiving any chemotherapy, physical therapy, or surgical treatment for ovarian lesions
* Wtih pathological ovarian results
* Willing to be tested and signed an informed consent form
* With available data of plasma CA125, Human epididymis protein 4 and effective imaging results

Exclusion Criteria:

* Not meeting all the including criteria
* WithoutoOvarian pathology or surgical pathology information could not be obtained
* A sample of patients withdrawing from the trial
* Samples that the investigator believes should be excluded from this trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pelvic mass or adnexal mass ready for surgical exploration
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity | One month
  Diagnostic sensitivity of methylation assay for detecting epithelial ovarian cancer
Diagnostic specificity | One month
  Diagnostic specificity of methylation assay for detecting epithelial ovarian cancer

SECONDARY OUTCOMES:
Progression-free survival | Two years
  Progression-free survival after the last treatment for cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China